CLINICAL TRIAL: NCT07325305
Title: The PROTECT Trial Physical Activity and Exercise During Early Treatment for Children With Acute Lymphoblastic Leukaemia to Protect Against Sarcopenia and Improve Frailty Outcomes: a Pilot Randomised Controlled Trial
Brief Title: Physical Activity and Exercise During Early Treatment Phases for Childhood Acute Lymphoblastic Leukaemia to Protect Against Muscle Loss and Improve Frailty Outcomes
Acronym: PROTECT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025/ETH01569
Record Dates: First submitted 2025-12-18; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenia; Acute Lymphoblastic Leukemia
Keywords: exercise; physical activity; behaviour change; paediatrics
MeSH Terms: conditions — Sarcopenia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Motor Activity | interventions — Exercise; Wearable Electronic Devices

STUDY DESIGN:
Intervention Model Description: Cohort observational study with embedded randomised control trial with randomisation 1:1 ratio to intervention and control group for those identified with sarcopenia after induction phase of treatment for acute lymphoblastic leukaemia.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention the provider of the intervention will not be blinded and nor will the participant. The investigator will be blinded where possible and any unblinding will be recorded and reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Observation cohort (No Intervention): These participants did not have early signs of sarcopenia at the post induction therapy assessment point, but will be followed up at all timepoints to better understand the natural progression of acute lymphoblastic leukaemia.
  Usual care is a ward based physiotherapist service which is reactive and referral based only.
- Usual care control group (No Intervention): These participants demonstrated early signs of sarcopenia at the post induction phase of treatment assessment point and were randomised to the control group. Usual care is a ward based physiotherapist service which is reactive and referral based only.
- Intervention group (Experimental): These participants demonstrated early signs of sarcopenia at the post induction phase of treatment assessment point and were randomised to the intervention group. The intervention group receives 9 weeks of goal setting and physical activity behaviour change coaching, as well as concurrently receiving 8 weeks of structured exercise sessions weekly (45-60 minutes per session x 3/week). These sessions are individualised based on the participant's functional performance outcomes from the assessment prior to randomisation, with a resistance strength training and progressive overload principles. The delivery of the specific exercises will be based on a pragmatic, participation based focus and will incorporate the individual's development stage, age, interests and enjoyment.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — These participants demonstrated early signs of sarcopenia at the post induction phase of treatment assessment point and were randomised to the intervention group. The intervention group receives 9 weeks of goal setting and physical activity behaviour change coaching (with activity tracking via Fitbit for continuous feedback) as well as concurrent 8 weeks of 3x45-60 minute structured exercise sessions weekly. These are individualised based on their functional performance outcomes from the assessment prior to randomisation with a resistance strength training and progressive overload principles. The delivery of the specific exercises will be based on a pragmatic, participation based focus and will incorporate the individuals development stage, age, interests and enjoyment.
  Other Names: physical activity; behaviour change; wearable device
  Arms: Intervention group

SUMMARY:
This is a small trial testing out a new approach before doing a bigger study. Researchers are observing a group of children/adolescents (ages 5-17) with acute lymphoblastic leukemia (ALL) and testing a physical activity and exercise program on a group of them who after 5 weeks of treatment show signs of weakness or frailty.

Kids who are NOT losing muscle aren't part of the exercise trial - they're just monitored over time to see how they do.

The goal:

To see if an exercise program helps kids who are getting weaker from acute lymphoblastic leukemia treatment build back/maintain their strength, compared to kids who don't do the extra intervention. The study will also look at if this way of measuring muscle weakness works well for kids with cancer.

DETAILED DESCRIPTION:
This is a pilot randomised controlled trial with a hybrid implementation design. At 5 weeks following an acute lymphoblastic leukaemia diagnosis children/adolescents (5-17 years) will be assessed for frailty using a novel frailty framework, to evaluate their frailty risk and identify those with signs of sarcopenia.

Children with signs of sarcopenia will be randomised to one of two groups:

1. Standard care only, or,
2. Physical activity and strengthening intervention plus activity tracking with a Fitbit (A wearable electronic activity tracker) This study will evaluate if the implementability of this intervention as well as the limited efficacy and investigate the framework for frailty used in this study.

It is known that children undergoing acute treatment for ALL experience signs of frailty from as early as 6 weeks post diagnosis. It is known that physical activity and exercise is safe and effective for children though it is most commonly conducted as a reactive therapy when children have already significantly deteriorated.

Very little is known regarding the pathophysiology that drives sarcopenia in children with cancer and there are no standardised diagnostic criteria, assessment tools or treatments. Often studies limit diagnosis to muscle ultrasound alone, omitting functional assessment. It has been recommended that a standardised criteria incorporating muscle mass (by ultrasound) and functional measurements (such as hand grip strength), should be established. This study aims to create a frailty framework including sarcopenia assessment ("muscle strength" and muscle mass "loss of muscle") as well as "slowness", "poor endurance", "low physical activity" as described in the outcome measurement section. This should contribute to a standardised criteria for sarcopenia as well as a criteria for identifying early signs of frailty with cut-offs.

The intervention aims to prevent frailty for participants with early signs of sarcopenia and currently there are no interventions that target frailty directly in children with cancer nor has frailty been investigated in the acute treatment phases of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5-17 years at the time of consent
* New diagnosis of acute lymphoblastic leukaemia <7 days
* Is planned to receive management for their cancer treatment at the trial site for the duration of the trial period
* Has a legally acceptable representative capable of understanding the informed consent document in English and providing consent on the participant's behalf
* Have a family electronic device that can be linked with the tool to be used (Fitbit)

Exclusion Criteria:

* none

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-17 (Estimated); Primary Completion 2028-07-17 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with low muscle mass on muscle ultrasound at 16 weeks | Baseline, 16 weeks
  Low muscle mass is defined as a 10% reduction on ultrasound in the cross-sectional area rectus femoris when comparing the ultrasound at enrolment/diagnosis with the ultrasound post intervention (prior to delayed intensification).
Mean change between-groups at 16 weeks in grip strength with handheld dynamometry | Baseline, 16 weeks
  Low muscle strength is defined as reduced grip strength with handheld dynamometry, where results are 2 standard deviations (SD) below normal with reference to age specific z scores
Mean change between-groups at 16 weeks in knee extension hand held dynamometry | Baseline, 16 weeks
  Low muscle strength is defined as reduced knee extension, where results are 2 standard deviations below normal with reference to age specific z scores.
Proportion of participants with low lean muscle mass on Dual-Energy X-ray Absorptiometry (DEXA) scan at 16 weeks | 5 weeks and 16 weeks
  <1.5 SD age specific z scores DEXA scan
Mean change of participants with low lean muscle mass on DEXA at 16 weeks | 5 weeks, 16 weeks and 24 weeks
  <1.5 SD age specific z score for lean muscle mass on DEXA scan
Acceptability measured by Theoretical Framework of Acceptability (TFA) survey | Baseline, mid intervention (4-7 weeks), 16 weeks (post intervention)
  The TFA is a generic survey specifically altered for the PROTECT study with 9 questions scoring 1-5. A score of 36 or higher is considered acceptable.
Qualitative acceptability | 16 weeks
  Measured by a semi-structured interview designed with Theoretical Domains Framework (TDF) and TFA theory
Fidelity of the intervention | Post-randomisation through to the final intervention session [anticipated at 15 weeks]
  proportion of completed intervention components of those offered and delivered
Feasibility of the intervention measured by the attrition rate | through study completion, approximately 17 months
  rate of attrition of participants from the trial
Feasibility of the intervention measured by screening rate | through study completion, approximately 17 months
  number of participants screened by the research team compared to number of eligible children admitted to ward across the study period.
Satisfaction of participants during the intervention | Post-randomisation through to the final intervention session [anticipated at 15 weeks]
  Using a Smiley face likert scale (5-point scale) of enjoyment, the children will be asked to rate their satisfaction following the completion of the intervention. A score of 4 or more is considered 'enjoyed'.

SECONDARY OUTCOMES:
Mean change in low Lumbar spine bone mineral density measured by DEXA | 5 weeks, 16 weeks and 24 weeks
  change over time to Lumbar spine bone mineral density, low is considered <1.5 SD of weight and age z-scores
Mean change in steps per day from 5 weeks to 16 weeks and Final visit | 5 weeks, 16 weeks, 24 weeks
  Measured using the Fitbit Inspire 3 for a 7 day period at week 5, week 16 and end of trial time points
Mean change in subjective Muscle Strength measured via the Patient-Reported Outcomes Measurement Information System (PROMIS) | 5 weeks, 16 weeks and 24 weeks
  subjective muscle strength survey comparing change in overall score from 5 weeks, 16 weeks and end of trial
Mean change in subjective Frailty measured via the Ped-SARC-F (Paediatric, Strength, Assistance with walking, Rising from a chair, Climbing stairs, and Falls): subjective sarcopenia questionnaire | 5 weeks, 16 weeks and 24 weeks
  The PED-SARC-F is a screening tool used to identify sarcopenia in pediatric patients, particularly those undergoing hemato-oncology treatment. The PED-SARC-F is a child-specific version of the standard SARC-F questionnaire used to assess sarcopenia in adults.
Proportion of participants with malnutrition measured by Malnutrition Score | 5 weeks, 16 weeks and 24 weeks
  The malnutrition score identifies the presence and severity of malnutrition based on z scores for weight-for-height/length
Mean change between-groups at 16 weeks in tibialis anterior strength with handheld dynamometry | Baseline, 16 weeks
  Low muscle strength is defined as reduced tibialis anterior strength with handheld dynamometry, where results are 2 standard deviations below normal with reference to age specific z scores.
Proportion of participants with low lower limb power evaluated by Jump Forward | 5 weeks, 16 weeks and 24 weeks
  Low lower limb power is defined by a Long jump distance <1.5 SD from age related z scores. Long jump is measuring the furthest horizontal distance jumped from a standing start. The assessment will be completed in line with standardised procedures.
Mean change in lower limb endurance as measured by the 30 second chair stand | 5 weeks, 16 weeks and 24 weeks
  Lower limb endurance is measured by the number of stands (established as full hip and knee extension) achieved in 30 seconds. The assessment will be completed in line with the standardised procedures. Change will be measured over time.
Proportion of participants with low lower limb endurance as measured by the 30 second chair stand | 5 weeks, 16 weeks and 24 weeks
  Low lower limb endurance is defined by <1.5 SD from the age related z scores in the 30 second chair stand which measures number of stands from a chair completed in 30 seconds.
Mean change in upper limb endurance as measured by the 30 second timed push ups | 5 weeks, 16 weeks and 24 weeks
  Upper limb endurance is measured by the number of knee push ups a participant can complete in 30 seconds. This assessment will be carried out in-line with the standardised sub-section of the Bruininks-Oseretsky Test of Motor Proficiency, 2nd Edition (BOT-2).
Proportion of participants with low upper limb endurance evaluated by the 30 second timed push up | 5 weeks, 16 weeks and 24 weeks
  low upper limb endurance is defined as <1.5 SD from age related z scores in the 30 second timed push up test (the number of knee push ups a participant can complete in 30 seconds).This assessment will be carried out in-line with the standardised sub-section of the Bruininks-Oseretsky Test of Motor Proficiency, 2nd Edition (BOT-2).
mean change in mobility as assessed by the 10 meter walk run test | 5 weeks, 16 weeks and 24 weeks
  Mobility is assessed using the 10-meter walk/run test (10MWRT). This is a timed test that measures walking or running speed over a 10m distance. It's used to assess mobility, gait, and balance. The assessment will be completed in line with the standardised procedures.
Proportion of participants with low mobility evaluated by the 10 meter walk run test | 5 weeks, 16 weeks and 24 weeks
  Low mobility is considered <1.5 SD of age related Z scores for the 10-meter walk/run test (10MWRT). This is a timed test that measures walking or running speed over a 10m distance. It's used to assess mobility, gait, and balance. The assessment will be completed in line with the standardised procedures.
Mean change in mobility endurance evaluated by the 100 meter walk run test | 5 weeks, 16 weeks, 24 weeks
  Mobility endurance is assessed using the 100-meter walk/run test (10MWRT). This is a timed test that measures walking or running speed over a 100m distance. It's used to assess mobility, gait, and balance. The assessment will be completed in line with the standardised procedures.
Proportion of participants with low mobility endurance evaluated by the 100 meter walk run test | 5 weeks, 16 weeks, 24 weeks
  Low mobility endurance is considered <1.5 SD of age related Z scores for the 100-meter walk/run test (100MWRT). This is a timed test that measures walking or running speed over a 100m distance. It's used to assess mobility, gait, and balance. The assessment will be completed in line with the standardised procedures.
Mean change for ability to climb stairs as measured by the Timed Up and Down Stairs (TUDS) | 5 weeks, 16 weeks and 24 weeks
  Ability to climb stairs will be measured using the timed stairs test which will be conducted on a set of 13 stairs with handrails. The time taken to walk up the stairs, turn around, and walk back down as quickly as possible was recorded. The assessment will be completed in line with the standardised procedures.
Proportion of participants with low ability to climb stairs evaluated by the Timed Up and Down Stairs (TUDS) | 5 weeks, 16 weeks and 24 weeks
  Low ability to climb stairs will be defined as <1.5 SD from age related z scores for the timed stairs test which will be conducted on a set of 13 stairs with handrails. The time taken to walk up the stairs, turn around, and walk back down as quickly as possible was recorded. The assessment will be completed in line with the standardised procedures.
Mean change in ability to rise from the floor as measured by the Time Rise from Floor | 5 weeks, 16 weeks and 24 weeks
  Ability to rise from floor is measured by the Timed rise from floor test which is conducted starting in supine and timed to stand with a graded quality assessment. The test will be conducted in line with standardised procedures.
Proportion of participants with low ability to rise from the floor evaluated by the timed rise from floor test | 5 weeks, 16 weeks, 24 weeks
  Low ability to rise from floor is defined as <1.5 SD from age related z scores in the Timed rise from floor test which is conducted starting in supine and timed to stand with a graded quality assessment. The test will be conducted in line with standardised procedures.
Mean change in ability to hop forwards as evaluated by the 6 meter hop test | 5 weeks, 16 weeks and 24 weeks
  Ability to hop is measured by 6 meter Hop forwards will be assessed as the furthest horizontal distance hopped from a standing start, and fasted hopping speed over 6 metres. Completed each side. The assessment will be completed in-line with standardised procedures
Proportion of participants with low ability to hop evaluated by the 6m hop test | 5 weeks, 16 weeks and 24 weeks
  low ability to hop forwards is defined as <1.5 SD from the age related Z scores of the 6m hop forward test.
  Hop forwards will be assessed as the furthest horizontal distance hopped from a standing start, and fasted hopping speed over 6 metres. Completed each side. The assessment will be completed in-line with standardised procedures
Proportion of chemotherapy induced peripheral neuropathy as measured by the Paediatric modified total neuropathy score | 5 weeks, 16 weeks and 24 weeks
  A score of >4 /32 is considered chemotherapy induced peripheral neuropathy on the paediatric modified total neuropathy score assessment. This is a standardised assessment combining subjective and objective elements, resulting in a score that indicates severity of a neuropathy. Assessment will be carried out according to standard procedure
Mean change in subjective fatigue evaluated by the PROMIS-Fatigue module questionnaire | 5 weeks, 16 weeks, 24 weeks
  PROMIS is a set of person-centred measures that evaluates and monitors physical, mental, and social health in children. The PROMIS measures across several health domains. Each domain takes ~ 3 min to complete. Within PROTECT we will use the parent proxy (age 5-17) and Pediatric (age 8-17
Mean change in subjective pain experience evaluated by the PROMIS-pain interference and behaviour module questionnaire | 5 weeks, 16 weeks and 24 weeks
  PROMIS is a set of person-centred measures that evaluates and monitors physical, mental, and social health in children. The PROMIS measures across several health domains. Each domain takes ~ 3 min to complete. Within PROTECT we will use the parent proxy (age 5-17) and Pediatric (age 8-17
Mean change in subjective sleep impairment evaluated by the PROMIS-sleep disturbance and impairment module questionnaire | 5 weeks, 16 weeks and 24 weeks
  PROMIS is a set of person-centred measures that evaluates and monitors physical, mental, and social health in children. The PROMIS measures across several health domains. Each domain takes ~ 3 min to complete. Within PROTECT we will use the parent proxy (age 5-17) and Pediatric (age 8-17
Mean change in subjective strength evaluated by the PROMIS-Strength impact questionnaire | 5 weeks, 16 weeks, 24 weeks
  PROMIS is a set of person-centred measures that evaluates and monitors physical, mental, and social health in children. The PROMIS measures across several health domains. Each domain takes ~ 3 min to complete. Within PROTECT we will use the parent proxy (age 5-17) and Pediatric (age 8-17
Mean change in subjective stress evaluated by the PROMIS-psychological stress questionnaire | 5 weeks, 16 weeks and 24 weeks
  PROMIS is a set of person-centred measures that evaluates and monitors physical, mental, and social health in children. The PROMIS measures across several health domains. Each domain takes ~ 3 min to complete. Within PROTECT we will use the parent proxy (age 5-17) and Pediatric (age 8-17

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Conyers, A/Prof Paediatric Oncologist, Study Director — Murdoch Children's Research Institute, Royal Children's Hospital (Melbourne), University of Melbourne
Locations (1):
- Royal Children's Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
There is an optional consent for the data collected to be used in future studies however, there are no data sharing agreements in place and therefore future studies would be using data under the original data agreements and protocols. A protocol publication is planned and will be linked to the registration when it is complete.